CLINICAL TRIAL: NCT04524650
Title: Construction and Evaluation of the Early Identification for Oxaliplatin Induced Portal Hypertension
Brief Title: Early Diagnosis of Oxaliplatin-induced Portal Hypertension
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Shiyao Chen, Professor, Shanghai Zhongshan Hospital
Other Study IDs: PLAEGV-DIA
Record Dates: First submitted 2020-08-20; First posted 2020-08-24 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Gastroesophageal Varices; Colorectal Cancer; Received Oxaliplatin-based Chemotherapy
Keywords: portal hypertension; splenomegaly; colorectal carcinoma; oxaliplatin; hepatotoxicity
MeSH Terms: conditions — Colorectal Neoplasms; Hypertension, Portal; Splenomegaly

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- stage 0: without liver function injury or splenomegaly
  Interventions: Diagnostic Test: the level of vWF
- stage 1: occurrence of liver function injury (ALT or AST > 2 ULN (upper limit of normal)
  Interventions: Diagnostic Test: the level of vWF
- stage 2: occurrence of splenomegaly or reduced platelet count (<150 X10^9/L)
  Interventions: Diagnostic Test: the level of vWF
- stage 3: occurrence of portal hypertension and/or gastroesophageal varices
  Interventions: Diagnostic Test: the level of vWF

INTERVENTIONS:
Diagnostic Test: the level of vWF — the peripheral level of vWF

SUMMARY:
Oxaliplatin has been used as the first choice for the adjuvant chemotherapy of colorectal cancer and it has significantly improved the outcomes in patients with colorectal cancer. However, hepatotoxicity is the potentially problematic adverse effect of oxaliplatin. The pathological evaluation of non-tumoral liver from patients with advanced colorectal cancer undergoing neoadjuvant oxaliplatin-based treatment has provided histological evidence of hepatic sinusoidal injury. Oxaliplatin-induced sinusoidal injury can persist for more than 1 year after the completion of chemotherapy, and the increase in splenic volume may be a predictor of irreversible sinusoidal damage. In this current study, the investigators aim to evaluate the values of potential biomarkers in diagnosing patients with oxaliplatin-induced gastroesophageal varices after colorectal cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18-75
* Had a history of oxaliplatin-based chemotherapy for the treatment of colorectal cancer surgery;

Exclusion Criteria:

* Combined known etiologies of chronic liver disease, including hepatitis, primary biliary cirrhosis, schistosomiasis, and non-alcoholic fatty liver disease.
* With colorectal cancer required further anti-tumor treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had a history of colorectal cancer and received oxaliplatin-based chemotherapy
Sampling Method: Probability Sample
Enrollment: 370 (Estimated)
Dates: Start 2020-08-31 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
the severity of portal hypertension | 1 day (the same time as diagnosis)
  High portal pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology and Hepatology, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Huang X, Li F, Wang L, Xiao M, Ni L, Jiang S, Ji Y, Zhang C, Zhang W, Wang J, Chen S. Endoscopic treatment of gastroesophageal variceal bleeding after oxaliplatin-based chemotherapy in patients with colorectal cancer. Endoscopy. 2020 Sep;52(9):727-735. doi: 10.1055/a-1157-8611. Epub 2020 May 7. PMID 32380558
- [Result] Aloia T, Sebagh M, Plasse M, Karam V, Levi F, Giacchetti S, Azoulay D, Bismuth H, Castaing D, Adam R. Liver histology and surgical outcomes after preoperative chemotherapy with fluorouracil plus oxaliplatin in colorectal cancer liver metastases. J Clin Oncol. 2006 Nov 1;24(31):4983-90. doi: 10.1200/JCO.2006.05.8156. PMID 17075116